CLINICAL TRIAL: NCT05960162
Title: Role of 90K/Mac-2 BP as an Indicator of Early Response to Infliximab Therapy in IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsattar Mohammed Madani, assistant lecturer of internal medicine, Assiut University
Other Study IDs: 04-2023-100093
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 90K — Blood test

SUMMARY:
The aim of this study is to analyze the relationship between 90K serum levels measured at baseline and after induction in IBD patient undergoing infliximab therapy, in order to clarify the role of serum 90K as an adjuvant biomarker for IBD patients in the active phase. Furthermore, the study aims to evaluate the clinical usefulness of this new biomarker in the management of IBD patients undergoing infliximab therapy.

DETAILED DESCRIPTION:
Type of the Study: The current work will be single cohort study.

Study settings: IBD outpatient clinic at Rajhy gastroenterology and Hepatology Hospital at Assiut University Hospital.

Study Duration: June 2023- June 2024 Study population: Participants will be 50 patients were recently diagnosed with Inflammatory Bowel Disease (IBD), Crohn's disease (CD) and Ulcerative Colitis (UC), undergoing the anti-TNF drug infliximab. Infliximab therapy will be administered intravenously initially at a dose of 5 mg/kg/ dose, and then after two and six weeks after the first dose, and fulfill the following inclusion criteria

Inclusion Criteria:

1. Adult male and female patients aged 18-60 years old.
2. IBD patients, diagnosis was confirmed by biopsy and histopathology, scheduled for treatment with anti-TNF therapy, Infliximab, and no previous treatment with anti-TNF therapy.

Exclusion Criteria:

1. Comorbidities (assessed with the Charlson Comorbidity Index).
2. Ongoing immunosuppressive or immunomodulatory therapy.
3. A malignant neoplasm in the last 10 years.
4. Pregnancy or breast feeding.
5. The need for artificial nutrition.

Study assay:

1. History taking and clinical examination, including the time and duration of diagnosis, manifestations of disease severity, and previous treatment received.
2. Laboratory investigations:

A. Routine investigations: such as complete blood count, liver function test (including serum albumin, liver enzymes, bilirubin), kidney function test (serum urea and creatinine, GFR), ESR and C - reactive protein.

B. The concentration of serum 90K glycoprotein is determined by ELISA assay, according to the manufacturer's instruction. Serum levels will be withdrawn before the first dose and after the third dose.

Statistical Tests:

Statistical tests will be performed with frequency and cross tabulations for categorical variables. Data will be reported as Mean+/- Standard Deviation (M +/- SD) for all numerical variables.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients aged 18-60 years old.
2. IBD patients, diagnosis was confirmed by biopsy and histopathology, scheduled for treatment with anti-TNF therapy, Infliximab, and no previous treatment with anti-TNF therapy.

Exclusion Criteria:

* 1. Comorbidities (assessed with the Charlson Comorbidity Index). 2. Ongoing immunosuppressive or immunomodulatory therapy. 3. A malignant neoplasm in the last 10 years. 4. Pregnancy or breast feeding. 5. The need for artificial nutrition.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be 50 patients were recently diagnosed with Inflammatory Bowel Disease (IBD), Crohn's disease (CD) and Ulcerative Colitis (UC), undergoing the anti-TNF drug infliximab. Infliximab therapy will be administered intravenously initially at a dose of 5 mg/kg/ dose, and then after two and six weeks after the first dose, and fulfill the following inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-17 (Estimated)

PRIMARY OUTCOMES:
evaluate the clinical usefulness of this new biomarker in the | 12 months

IPD SHARING:
Plan to Share IPD: Undecided